CLINICAL TRIAL: NCT01393717
Title: A Phase II Study of Brentuximab Vedotin as Salvage Therapy for Hodgkin Lymphoma Prior to Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Brentuximab Vedotin Before Autologous Stem Cell Transplant in Treating Patients With Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11051; NCI-2011-01135 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-07-08; First posted 2011-07-13 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Recurrent Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (brentuximab vedotin) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses. Patients in the new cohort receive regular study dose of brentuximab vedotin for courses 1 and 2. Patients not achieving CR after 2 courses receive higher-dose brentuximab vedotin IV over 60 minutes on day 1 for 2 additional courses.
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — Given IV
  Other Names: anti-CD30 ADC SGN-35; anti-CD30 antibody-drug conjugate SGN-35; antibody-drug conjugate SGN-35; SGN-35; Adcetris

SUMMARY:
This phase II trial studies how well brentuximab vedotin before autologous (taken from an individual's own cells) stem cell transplant works in treating patients with Hodgkin lymphoma. Monoclonal antibody-drug conjugates, such as brentuximab vedotin, can block cancer growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this study is to determine the activity of salvage brentuximab vedotin in Hodgkin lymphoma prior to autologous hematopoietic stem cell transplantation, as measured by overall response rate (ORR).

SECONDARY OBJECTIVES:

I. To describe the safety, toxicity, and tolerability of brentuximab vedotin as a salvage regimen.

II. To summarize the stem cell mobilization results of patients receiving brentuximab vedotin as salvage therapy (e.g., total cluster of differentiation (CD)34+ cell yield, number of apheresis days, proportion of patients who achieve >= 3 x 10^6 CD34+ cells/kg).

III. To evaluate potential changes in Hodgkin lymphoma biological markers of patients treated with brentuximab vedotin as first line salvage therapy.

IV. To examine and characterize the outcomes of patients who receive brentuximab vedotin as first line salvage followed by autologous hematopoietic stem cell transplantation (AHCT) (e.g., toxicity, 2-year progression free survival [PFS], overall survival [OS], relapse-progression incidence and non-relapse mortality rate [NRM])

OUTLINE:

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses.

Patients in the new cohort receive regular study dose of brentuximab vedotin for courses 1 and 2. Patients not achieving complete remission (CR) after 2 courses receive higher-dose brentuximab vedotin IV over 60 minutes on day 1 for 2 additional courses.

After completion of study treatment, patients are followed up at 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented or cytologically confirmed Hodgkin lymphoma with CD 30 expression
* Patients must have absolute neutrophil count (ANC) >= 1000/uL; neupogen (filgrastim) can be given prior to start of SGN-35 (brentuximab vedotin) and during SGN-35 treatment to achieve target ANC >= 1000/uL
* Patients must have platelets (Plts) >= 50,000/uL; platelet transfusion can be given prior to the start of SGN-35 and during SGN-35 treatment to achieve a target plt >= 50,000/uL
* Patients must have measurable disease > 1.5 cm evidenced by computed tomography (CT) scan of the neck/chest/abdomen(abd)/pelvis or CT/positron emission tomography (PET) scans
* Patient must be either primary refractory to one frontline induction therapy or relapsed after one frontline induction therapy; patients who do not achieve complete remission after induction therapy are also eligible
* Patients cannot have had a second line salvage treatment (chemotherapy, biologic agents, investigational drugs, or radiation) or have had an autologous or allogeneic hematopoietic stem cell transplantation; patients can have had mixed frontline therapy such as 2-4 cycles of ABVD (doxorubicin, bleomycin, vinblastine and dacarbazine) followed by 2-4 cycles of bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPP) as long as the induction chemotherapy is not more than 8 cycles in total length
* Radiation use as part of induction regimen or consolidation (within 90 days after completion of induction chemotherapy) is allowed
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male subject agrees to use an acceptable method of contraception for the duration of the study
* Life expectancy of greater than 3 months
* Karnofsky performance status of > 60%
* ANC >= 1000/uL
* Plts >= 50,000/uL
* Total bilirubin within 1.5 x of the upper limit of normal (ULN) institutional limits, patients with elevation of unconjugated bilirubin alone, as in Gilbert's disease, are eligible
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 X institutional ULN (unless demonstrated Hodgkin lymphoma involvement of the liver)
* Calculated creatinine clearance >30 ml/min (unless demonstrated Hodgkin lymphoma involvement of the kidney)

ELIGIBILITY FOR 2.4 MG/KG DOSING IN THE NEW COHORT:

- In addition to the inclusion/exclusion criteria outlined, to be eligible for treatment with the higher 2.4 mg/kg dose of brentuximab vedotin in the new cohort of 20 additional patients, best response after 2 cycles of brentuximab vedotin administered at the 1.8 mg/kg dose, must be partial remission (PR) or stable disease (SD) as determined by radiographic imaging

Exclusion Criteria:

* Patient has > 1.5 x ULN total bilirubin, unless history of Gilbert's syndrome
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Patient has hypersensitivity to brentuximab vedotin
* Female subject is pregnant or breast-feeding; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patient has received other investigational drugs within 14 days before treatment of treatment with brentuximab vedotin
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Patients with other active malignancies (no evidence of other cancer or life expectancy greater than 5 years) are ineligible for this study
* Patients with active central nervous system (CNS) disease or history of brain metastases (mets) are excluded from study
* Patients may be on steroids prior to initiation of treatment as long as by cycle 1 day 1 steroids use was tapered down less than or equal to 20 mg of prednisone.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-10-20 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chen, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Weill Medical College, Cornell University, New York, New York

REFERENCES:
- [Derived] Herrera AF, Palmer J, Martin P, Armenian S, Tsai NC, Kennedy N, Sahebi F, Cao T, Budde LE, Mei M, Siddiqi T, Popplewell L, Rosen ST, Kwak LW, Nademanee A, Forman SJ, Chen R. Autologous stem-cell transplantation after second-line brentuximab vedotin in relapsed or refractory Hodgkin lymphoma. Ann Oncol. 2018 Mar 1;29(3):724-730. doi: 10.1093/annonc/mdx791. PMID 29272364
- [Derived] Chen R, Palmer JM, Martin P, Tsai N, Kim Y, Chen BT, Popplewell L, Siddiqi T, Thomas SH, Mott M, Sahebi F, Armenian S, Leonard J, Nademanee A, Forman SJ. Results of a Multicenter Phase II Trial of Brentuximab Vedotin as Second-Line Therapy before Autologous Transplantation in Relapsed/Refractory Hodgkin Lymphoma. Biol Blood Marrow Transplant. 2015 Dec;21(12):2136-2140. doi: 10.1016/j.bbmt.2015.07.018. Epub 2015 Jul 26. PMID 26211987

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort #1: Patients receive brentuximab vedotin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses.
- Cohort #2: Patients receive regular study dose of brentuximab vedotin for courses 1 and 2. Patients not achieving CR after 2 courses receive higher-dose brentuximab vedotin IV over 60 minutes on day 1 for 2 additional courses.
Period: Overall Study
Arm/Group | Cohort #1 | Cohort #2
Started | 37 | 20
Completed | 37 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Patients receive salvage brentuximab vedotin IV.
Arm/Group | All Study Participants
Number analyzed (Participants) | 57
Age, Continuous [Median (Full Range); unit: years] | 32 [11 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 36
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Among Patients With Salvage Brentuximab Vedotin (BV)
Description: The overall response rate is calculated as the percent of evaluable patients that have confirmed CR or PR by radiographic imaging, and the exact 95% confidence interval is calculated for this estimate. Per Revised Response Criteria for Malignant Lymphoma (Cheson et al. 2007) for target lesions and assessed by CT/PET scans: Complete Response (CR), complete disappearance of all detectable clinical and radiographic evidence of disease; Partial Response (PR), ≥50% decrease in the sum of the product of the diameters of up to six of the largest dominant nodes or nodal masses.
Time Frame: 21 days after completion of last course of study treatment, up to 5 years
Population: Among the 57 enrolled patients, only 56 patients were evaluable for efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Groups:
- Patients Receive Brentuximab Vedotin: Patients receive brentuximab vedotin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses. Patients in the new cohort receive regular study dose of brentuximab vedotin for courses 1 and 2. Patients not achieving CR after 2 courses receive higher-dose brentuximab vedotin IV over 60 minutes on day 1 for 2 additional courses.
Arm/Group | Patients Receive Brentuximab Vedotin
Number analyzed (Participants) | 56
percentage of participants with response | 75.0 [61.6 to 85.6]

2. Primary Outcome: Complete Response (CR) Rate Among Patients With Salvage Brentuximab Vedotin (BV)
Description: The CR rate is calculated as the percent of evaluable patients that have confirmed CR by radiographic imaging, and the exact 95% confidence interval is calculated for this estimate. Per Revised Response Criteria for Malignant Lymphoma (Cheson et al. 2007) for target lesions and assessed by CT/PET scans: Complete Response (CR), complete disappearance of all detectable clinical and radiographic evidence of disease.
Time Frame: 21 days after completion of last course of study treatment, up to 5 years
Population: Among the 57 enrolled patients, only 56 patients were evaluable for efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | Patients Receive Brentuximab Vedotin
Number analyzed (Participants) | 56
percentage of participants with response | 42.9 [29.7 to 56.8]

3. Primary Outcome: Overall Response Rate in Cohort #2
Description: as for outcome 1
Time Frame: 21 days after completion of last course of study treatment, up to 5 years
Population: Among the 20 enrolled patients in Cohort #2, all the 20 patients were evaluable for efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Groups:
- Patients in Cohort #2: Patients receive regular study dose of brentuximab vedotin for courses 1 and 2. Patients not achieving CR after 2 courses receive higher-dose brentuximab vedotin IV over 60 minutes on day 1 for 2 additional courses.
Arm/Group | Patients in Cohort #2
Number analyzed (Participants) | 20
percentage of participants with response | 85.0 [62.1 to 96.8]

4. Primary Outcome: Complete Response (CR) Rate in Cohort #2
Description: as for outcome 2
Time Frame: 21 days after completion of last course of study treatment, up to 5 years
Population: Among the 20 enrolled patients in Cohort #2, all the 20 patients were evaluable for efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | Patients in Cohort #2
Number analyzed (Participants) | 20
percentage of participants with response | 55.0 [31.5 to 76.9]

5. Secondary Outcome: Total CD34+ Cell Dose Among Patients Receiving Brentuximab Vedotin Followed by Autologous Hematopoietic Stem Cell Transplantation
Description: Among the patients receiving salvage Brentuximab Vedotin (BV) followed by Autologous Hematopoietic Stem Cell Transplantation (AutoHCT), their total CD34+ cell yield by stem cell mobilization.
Time Frame: 60 days after completion of last course of study treatment, up to conditioning regimens
Population: Among the 57 enrolled patients, 50 patients receive BV followed by AutoHCT, 32 in Cohort #1 and 18 in Cohort #2.
Measure: Median (Full Range); unit: x10^6 cells/kg
Arm/Group | Cohort #1 | Cohort #2
Number analyzed (Participants) | 32 | 18
x10^6 cells/kg | 6.0 [2.6 to 34.0] | 8.0 [2.8 to 30.5]

6. Secondary Outcome: Progression Free Survival at Year Two Among AutoHCT Patients With BV
Description: Progression Free Survival (PFS) defined as the time from first treatment day (post AHCT) until objective or symptomatic relapse or death as a result of lymphoma or acute toxicity of treatment. Assessed by Kaplan-Meier survival analysis and 95% confidence intervals will be calculated using Greenwood's formula.
Time Frame: Assessed for up to 5 years, at least half of the surviving participants followed 2+ years
Population: Among the 57 patients receiving BV, only 50 patients had undergone autologous transplants.
Measure: Number (95% Confidence Interval); unit: survival probability
Groups:
- Patients With BV Followed by AutoHCT: Patients that received brentuximab vedotin followed by autologous transplants.
Arm/Group | Patients With BV Followed by AutoHCT
Number analyzed (Participants) | 50
survival probability | 0.67 [0.52 to 0.78]

7. Secondary Outcome: Overall Survival at Year Two Among AutoHCT Patients With BV
Description: Overall Survival (OS) defined as the time from first treatment day (post AHCT) until death. Assessed by Kaplan-Meier survival analysis and 95% confidence intervals will be calculated using Greenwood's formula.
Time Frame: Assessed for up to 5 years, at least half of the surviving participants followed 2+ years
Population: Among the 57 patients receiving BV, only 50 patients had undergone autologous transplants.
Measure: Number (95% Confidence Interval); unit: survival probability
Groups:
- Patients Received BV Followed by AutoHCT: Patients that received brentuximab (BV) vedotin followed by autologous transplants
Arm/Group | Patients Received BV Followed by AutoHCT
Number analyzed (Participants) | 50
survival probability | 0.93 [0.80 to 0.98]

ADVERSE EVENTS:
Time Frame: Death was monitored from Day 0 up to Year 5. Serious and other adverse events were assessed after each cycle of treatment, up to 5 years.
Arm/Group | Cohort #1 | Cohort #2
All-Cause Mortality (participants affected / at risk) | 6/37 | 2/20
Serious Adverse Events (participants affected / at risk) | 4/37 | 0/20
Other Adverse Events (participants affected / at risk) | 37/37 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort #1 (N=37) | Cohort #2 (N=20)
Fever (General disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort #1 (N=37) | Cohort #2 (N=20)
Anemia (Blood and lymphatic system disorders) | 8 (9) | 5 (5)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 5 (5) | 3 (3)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (11) | 6 (7)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 3 (4)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 11 (11) | 5 (5)
Fever (General disorders) | 4 (4) | 4 (4)
Flu like symptoms (General disorders) | 3 (3) | 0 (0)
Gait disturbance (General disorders) | 3 (3) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 3 (5) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 6 (6) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 14 (15) | 9 (9)
Alkaline phosphatase increased (Investigations) | 4 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 17 (21) | 8 (9)
Blood bilirubin increased (Investigations) | 3 (4) | 0 (0)
Cholesterol high (Investigations) | 5 (5) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (4) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 5 (8) | 1 (1)
Platelet count decreased (Investigations) | 3 (4) | 1 (1)
Weight gain (Investigations) | 0 (0) | 2 (2)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 8 (10) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (6) | 5 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 12 (15) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5) | 5 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (4)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (17) | 7 (11)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (7)
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 (16) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (7) | 9 (12)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 9 (11) | 11 (15)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT01393717/Prot_SAP_000.pdf